CLINICAL TRIAL: NCT04713046
Title: A Phase I Clinical Trial Assessing the Safety, Feasibility and Immunologic Correlates of Allogeneic HPV-specific Cluster of Differentiation 4 (CD4)+ T Cells in Advanced HPV16-associated Malignancies
Brief Title: Safety and Efficacy of Allogeneic HPV-specific T Cells in Adults With Recurrent or Metastatic HPV16+ Cancers
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: PapiVax Biotech, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J21112; IRB00244082 (Other: JHM IRB)
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: HPV 16+ Recurrent or Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Randomized 1:1, 2-arm open-label trial
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Allogeneic bone marrow transplant (Experimental): non-myeloablative allogeneic bone marrow transplant (BMT) from a haploidentical relative after vaccination with a therapeutic HPV vaccine series.
  Interventions: Biological: Non-myeloablative allogeneic bone marrow transplant from related donors vaccinated against HPV16
- CD8-depleted donor lymphocyte infusion (DLI) per dose escalation scheme (Experimental): CD8-depleted donor lymphocyte infusion per dose escalation scheme from a haploidentical relative after vaccination with a therapeutic HPV vaccine series.
  Interventions: Biological: CD8 reduced peripheral blood cells taken from related donors vaccinated against HPV16

INTERVENTIONS:
Biological: CD8 reduced peripheral blood cells taken from related donors vaccinated against HPV16 — Patients will receive CD8+ T cell-depleted peripheral blood cells at one of three dose levels following cyclophosphamide: 1) 10^6 CD4+ cells/kg; 2) 5 x 10^6 CD4+ cells/kg; or 3) 10^7 CD4+ cells/kg of recipient ideal body weight.
  Arms: CD8-depleted donor lymphocyte infusion (DLI) per dose escalation scheme
Biological: Non-myeloablative allogeneic bone marrow transplant from related donors vaccinated against HPV16 — Standard dosing for bone marrow graft (target dose of 4 x 10^8 nucleated cells/kg) and if progression at Day 90, will receive dose level 1 for the CD8-depleted DLI (106 CD4+ cell/kg).
  Arms: Allogeneic bone marrow transplant

SUMMARY:
In this study, haploidentical relatives of a patient with recurrent or metastatic HPV 16-associated malignancy will be vaccinated with a therapeutic human papillomavirus (HPV) vaccine series to generate HPV-specific leukocytes. The cancer patient with recurrent or metastatic HPV16+ cancer will then be randomized to one of two arms: 1) non-myeloablative allogeneic bone marrow transplant or 2) cluster of differentiation 8 (CD8)-depleted donor lymphocyte infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Have pathologically confirmed incurable, locally recurrent or metastatic HPV16+ HNSCC
2. Male or female ≥ 18 years of age
3. Have an human leukocyte antigen (HLA) partially mismatched (haploidentical) related donor. Acceptable donors include first degree relatives (parent, child, or haploidentical sibling), half-siblings, or second degree relatives (aunt, uncle, cousin, niece, nephew). A patient who has inherited a recombinant haplotype from the parents is eligible if the donor shares at least 1 HLA antigen at each of the HLA-A, HLA-B, and HLA DR isotype (HLA-DR) loci.
4. Prior treatment with a platinum-containing regimen
5. Patients with an FDA-approved indication to receive an anti-programmed cell death protein-1 (PD-1) or anti-programmed death-ligand1 (PD-L1) monoclonal antibody must have received at least one cycle of this therapy prior to receiving treatment on this trial
6. Life expectancy ≥ 4 months at time of screening
7. Measurable disease using RECIST 1.1. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been documented in such lesions
8. Eastern Cooperative Oncology Group (ECOG) performance status of < 2 (see Appendix A).
9. Adequate organ function per the protocol, as defined below:

   * Left ventricular ejection fraction > 35% (within 30 days of eligibility screening)
   * Total bilirubin < 3.0 mg/dl unless from Gilbert disease
   * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 4 x institutional upper limit of normal
   * Serum creatinine < 3.0 mg/dl
10. Willing and able to provide written informed consent

Exclusion Criteria:

1. Disease that is suitable for local therapy administered with curative intent
2. Requires vasopressor or ventilator support
3. Received antithymocyte globulin or similar anti-T-cell antibody therapy ≤ 4 weeks prior to Cycle 1 Day 1
4. Diagnosis of immunodeficiency or is receiving systemic steroid therapy >10 mg/day of prednisone or equivalent, or any other form of immunosuppressive therapy within 7 days prior to Cycle 1 Day 1 of study treatment.
5. Active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
6. Active infection requiring systemic therapy
7. History of (non-infectious) pneumonitis that required steroids or current pneumonitis
8. Received any live vaccine for up to 30 days prior to enrollment.
9. Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer not associated with HPV16.
10. Pregnancy or breastfeeding: females of childbearing potential must have a negative serum pregnancy test.
11. Female of childbearing potential or male with a female partner of childbearing potential unwilling to use a highly effective method of contraception (abstinence is acceptable) for the course of the study through 120 days after the last study dose since the effects of this therapy on the developing human fetus are unknown.
12. Inability to comply with study procedures
13. Received chemotherapy or targeted small molecule therapy within 2 weeks of the first dose of cyclophosphamide. Subjects must have recovered (ie, grade ≤ 1 or at baseline) from adverse events (AEs) due to a previously administered agent. Subjects with grade ≤ 2 neuropathy or grade ≤ 2 alopecia are an exception to this criterion.
14. Received prior radiotherapy within 2 weeks of the first dose of cyclophosphamide. Subjects must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1- week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
15. Carcinomatous meningitis; and/or active CNS metastases, unless metastases are treated and stable and the subject does not require systemic steroids.
16. Known history of human immunodeficiency virus (HIV), known active hepatitis B virus (HBV; e.g., hepatitis B surface antigen [HBsAg] reactive), or hepatitis C virus (HCV; e.g., HCV ribonucleic acid [RNA] is detected)
17. Prior treatment with HPV T cells

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | 12 months
  Determine the safety of the two interventions in patients with recurrent or metastatic HPV16-associated cancer. Safety will be monitored for every patient and we will document and grade every adverse event using the NCI CTCAE version 5.0.
Maximum Tolerated Dose (MTD) of Allogeneic CD4+ T cell Infusion | 12 months
  Determine the maximum tolerated dose (in CD4+ cells/kg) of allogeneic CD4+ T cells infused after cyclophosphamide in patients with recurrent or metastatic HPV16-associated cancer. We will use three dose levels of allogeneic CD4+ T cells: 1) 10^6 CD4+ cells/kg; 2) 5 x 10^6 CD4+ cells/kg; 3) 10^7 CD4+ cells/kg of recipient ideal body weight. We will implement a Bayesian optimal interval design to find the MTD with an observation period of 42 days for treatment-related toxicities.

SECONDARY OUTCOMES:
Number of toxicities as assessed by the NCI CTCAE version 5.0 | 12 months
  Count the toxicities of allogeneic BMT and HPV-specific CD4+ T cells in patients with recurrent or metastatic HPV16-associated cancer. Toxicities of treatment will be formally assessed and scored using the Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.
Progression-free survival (PFS) of allogeneic CD4+ T cell Infusion and allogeneic BMT | 12 months
  PFS is defined as the date from transplantation to the date of relapse/progression, death from any cause or last follow-up, whichever comes first. Kaplan-Meier curve will be generated and PFS will be estimated along with 95% confidence intervals.
Overall survival (OS) of allogeneic CD4+ T cell Infusion and allogeneic BMT | 12 months
  OS is defined as the date from infusion or transplantation to the date of death from any cause or last follow-up. A Kaplan-Meier curve will be generated along with 95% confidence intervals.
Overall Response of allogeneic CD4+ T cell Infusion and allogeneic BMT | Up to 12 months
  Response will be defined as per the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) and will be evaluated at 2, 6 and 12 months after transplantation or infusion.
Incidence of acute graft versus host disease (GVHD) | 12 months
  Each patient will be monitored for acute GVHD and we will grade acute GVHD using the consensus conference clinical grading of acute GVHD.

CONTACTS AND LOCATIONS:
Overall Officials: Tanguy Seiwert, MD, Principal Investigator — Johns Hopkins Sidney Kimmel Comprehensive Cancer Center
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No